CLINICAL TRIAL: NCT00749749
Title: A Phase II, Randomized, Single-dose, Unblinded Study to Compare the Efficacy and Safety of the CollaRx Bupivacaine Implant With the ON-Q PainBuster Post-op Pain Relief System in Women Following Abdominal Hysterectomy
Brief Title: Efficacy and Safety of the CollaRx Bupivacaine Implant Compared to the ON-Q Painbuster Following Abdominal Hysterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innocoll (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INN-CB-005
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Pain, Postoperative
Keywords: Abdominal Hysterectomy; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine collagen sponge (Experimental): Three Bupivacaine sponges placed at different levels within the surgical cavity; one deep within the vault, one at the incision line in the peritoneum and one at the dermal incision line.
  Interventions: Drug: Bupivacaine Collagen Sponge (CollaRx Bupivacaine Implant)
- ON-ON-Q PainBuster Post-op Pain relief SystemQ system (Active Comparator): Insertion of the ON-Q system catheter into the deep subcutaneous space overlying the fascia.
  Interventions: Drug: ON-Q PainBuster Post-op Pain relief System

INTERVENTIONS:
Drug: Bupivacaine Collagen Sponge (CollaRx Bupivacaine Implant) — The bupivacaine collagen sponge contains 70mg Type I bovine collagen and 50mg bupivacaine hydrochloride
  Other Names: CollRx Bupivacaine Implant
  Arms: Bupivacaine collagen sponge
Drug: ON-Q PainBuster Post-op Pain relief System — 5 mL/hr per catheter of 0.25% bupivacaine (12.5 mg) for 72 hours(total dose 360 mL [900 mg])
  Arms: ON-ON-Q PainBuster Post-op Pain relief SystemQ system

SUMMARY:
The purpose of this study is to determine whether the CollaRx Bupivacaine Implant is safe and effective in reducing the amount of narcotic pain medication needed to control pain during the first 96 hours after abdominal hysterectomy when compared to the ON-Q PainBuster Post-op Pain Relief System.

DETAILED DESCRIPTION:
Hysterectomy is the second most common surgery among women in the United States (US). Abdominal hysterectomy surgery may be performed to treat benign tumors, such as fibroids, heavy periods, painful periods and chronic pelvic pain. The most common route for performing hysterectomy is through an incision in the abdominal wall; however, about 20% are performed vaginally.Laparoscopic assisted vaginal hysterectomy is performed when warranted.

Bupivacaine is a local anesthetic (pain medication) that has an established safety profile. Collagen is a protein that is found in all mammals. The CollaRx Bupivacaine implant is a thin flat sponge made out of collagen that comes from cattle tendons and contains bupivacaine. When inserted into a surgical site, the collagen breaks down and bupivacaine is released at the site but very little is absorbed into the blood stream. The high levels of bupivacaine at the surgical site may result in less pain for several days after surgery.

The ON Q system consists of 1 elastometric pump with a fill volume of 270 mL containing 0.25% bupivacaine; 1 soaker catheter measuring 12.5 cm in size; and a fill port, tubing, clamp, filter and flow restrictor. The pump provides positive pressure and is portable. It may be attached to the patient's dressing or placed in a carrying pouch. The catheter is inserted directly into the surgical wound providing a continuous flow of bupivacaine into the wound. A capillary flow restricting orifice located at the end of the tubing controls the flow rate.

This study will compare the total narcotic use in patients with the CollaRx Bupivacaine Implant with the total narcotic use in patients with the ON Q PainBuster Post op Pain Relief System after abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Must be a woman who is ≥ 18 and ≤ 75 years of age.
* Has a body mass index (BMI) > 19 and < 40 kg/m2.
* Has planned an elective total abdominal hysterectomy for reasons other than malignancies (such as uterine adenocarcinoma, cervical cancer or leiomyosarcoma) to be performed according to standard surgical technique using a standard incision and under general anesthesia with the following caveats:

  * Laparoscopic procedures or supraumbilical or Maylard incisions will not be allowed.
  * A nonlaparoscopic incision for benign nonhysterectomy gynecological procedures (such as myomectomy or adnexal surgery) is acceptable if the surgical indication is not to treat pelvic pain.
  * No concomitant vaginal procedures such as anterior and posterior colporrhaphy (A&P repairs) are allowed. An abdominal urethropexy and an incidental appendectomy will be allowed.
* Has a risk classification of I, II or III according to the American Society of Anesthesiologists (ASA).
* Is nonpregnant (negative pregnancy test at Screening and Day 0 before surgery) and nonlactating.
* Is free of other physical or mental conditions that, in the opinion of the Investigator, may confound quantification of postoperative pain resulting from the abdominal hysterectomy.
* Has the ability to read, understand and comply with the study procedures and the use of the pain scales; is deemed capable of operating a patient controlled analgesia (PCA) device; and is able to communicate meaningfully with the study staff.
* Must voluntarily sign and date an informed consent form (ICF), approved by an Institutional Review Board (IRB), prior to the conduct of any study specific procedures.
* Must be able to fluently speak and understand English and be able to provide meaningful written informed consent for the study.

Exclusion Criteria:

* Has known hypersensitivity to amide local anesthetics, opioids, bovine products or to inactive ingredients of the test article or reference product.
* Has cardiac arrhythmias or atrioventricular (AV) conduction disorders.
* Concomitantly uses other amide local anesthetics.
* Concomitantly uses antiarrhythmics (eg, amiodarone), propranolol or strong/moderate cytochrome P450 (CYP) 3A4 inhibitors or inducers (eg, macrolide antibiotics and grapefruit juice).
* Has used long acting analgesics within 24 hours of surgery. Short acting analgesics such as acetaminophen may be used on the day of surgery but are subject to preoperative restrictions for oral intake.
* Has used aspirin or aspirin containing products within 7 days of surgery. Aspirin at a dose of ≤ 325 mg is allowed for cardiovascular prophylaxis if the patient has been on a stable dose regimen for ≥ 30 days prior to Screening.
* Has undergone major surgery within 3 months of the scheduled hysterectomy.
* Requires the use of Seprafilm® or other absorbable adhesion barriers for the scheduled hysterectomy.
* Requires any additional surgical procedures either related or unrelated to the abdominal hysterectomy during the same hospitalization (except for the specific allowed procedures noted in the Inclusion Criteria).
* Is required to receive neuraxial (spinal or epidural) opioid analgesics during the surgery.
* Has known or suspected history of alcohol or drug abuse or misuse within 3 years of Screening or evidence of tolerance or physical dependency on opioid analgesics or sedative hypnotic medications.
* Has used opioids or tramadol on an extended daily basis (> 7 days) prior to surgery. Patients who, in the Investigator's opinion, are developing opioid tolerance are to be excluded.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-09-10; Primary Completion 2008-12-22 (Actual); Study Completion 2008-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Prior, Study Director — Innocoll
Locations (1):
- Visions Clinical Research, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cusack SL, Minkowitz HS, Kuss M, Jaros M, Hemsen L. A randomized, multicenter, pilot study comparing the efficacy and safety of a bupivacaine-collagen implant (XaraColl((R))) with the ON-Q PainBuster((R)) Post-op Pain Relief System following open gynecological surgery. J Pain Res. 2012;5:453-61. doi: 10.2147/JPR.S37310. Epub 2012 Nov 2. PMID 23152696

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (11.50) | 43.4 (41.0) | 43.3 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Amount of Opioid Rescue Analgesia Used
Description: Higher value means worse outcome - Higher number reflects a need for more analgesia - For the first 24 hours after surgery, patients received IV morphine via a PCA pump as rescue analgesia. Patient demand for morphine was recorded. Measurement recorded in total Morphine Milligrams
Time Frame: 0 to 24 hours postoperatively
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: Morphine Milligrams
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System
Number analyzed (Participants) | 14 | 13
Morphine Milligrams | 46.85 (21.57) | 67.03 (32.416)

2. Secondary Outcome: Total Amount of Opioid Rescue Analgesia Used
Description: Higher score means worse outcome - Higher number means more Analgesia was needed. For the first 24 hours after surgery, patients received IV morphine via a PCA pump as rescue analgesia. Patient demand for morphine was recorded. After 24 hours, patients were offered hydrocodone/acetaminophen (maximum could not exceed 8 tablets per 24 hours of the 5/500 mg tablets [40 mg hydrocodone and 4000 mg acetaminophen]) or similar medication as determined by the Investigator for pain until discharge. If oral medication was insufficient for control of pain, IM or IV morphine could be administered.
Time Frame: 0 to 48 hours postoperatively
Population: ITT population
Measure: Mean (Standard Deviation); unit: Morphine equivalents
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System
Number analyzed (Participants) | 14 | 13
Morphine equivalents | 55.43 (22.770) | 74.85 (35.381)

3. Secondary Outcome: The Total Amount of Opioid Rescue Analgesia Used
Description: Higher score means worse outcome. Higher number means more Analgesia was needed. For the first 24 hours after surgery, patients received IV morphine via a PCA pump as rescue analgesia. Patient demand for morphine was recorded. After 24 hours, patients were offered hydrocodone/acetaminophen (maximum could not exceed 8 tablets per 24 hours of the 5/500 mg tablets [40 mg hydrocodone and 4000 mg acetaminophen]) or similar medication as determined by the Investigator for pain until discharge. If oral medication was insufficient for control of pain, IM or IV morphine could be administered.
Time Frame: 0 to 96 hours postoperatively
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Morphine equivalents
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System
Number analyzed (Participants) | 14 | 13
Morphine equivalents | 67.87 (28.175) | 90.77 (46.114)

4. Secondary Outcome: Total Use of Opioid Rescue Analgesia (mg) Over 0 to 72 Hours
Description: as for outcome 3
Time Frame: 0 to 72 Hours
Population: ITT population
Measure: Mean (Standard Deviation); unit: Morphine equivalents
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System
Number analyzed (Participants) | 14 | 13
Morphine equivalents | 61.98 (25.27) | 85.36 (41.887)

5. Secondary Outcome: Time to First Use of Opioid Rescue Analgesia
Description: Higher score has a better outcome
Time Frame: 0 to 72 hours
Population: Intent-to-Treat Population
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System
Number analyzed (Participants) | 14 | 13
Hours | 0.78 [0.43 to 1.02] | 0.57 [0.33 to 0.58]

6. Secondary Outcome: VAS Pain Intensity Scores Over Time AT REST
Description: For the VAS assessment, patients measured their pain intensity at rest using a horizontal 100-mm VAS scale labeled as follows: No Pain (0 mm) as the left anchor and Worst Pain Imaginable (100 mm) as the right anchor.
Time Frame: Hour 1, 1.5, 2,3,6,9,12,18,24,36,48,72,96
Population: ITT population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System
Number analyzed (Participants) | 14 | 13
units on a scale
  Hour 1.0 | 75.2 (21.32) | 74.5 (22.75)
  Hour 1.5 | 66.3 (24.96) | 66.5 (28.65)
  Hour 2 | 61.5 (26.92) | 68.6 (26.52)
  Hour 3 | 52.2 (21.71) | 60.9 (29.85)
  Hour 6 | 49.9 (32.15) | 45.8 (24.49)
  Hour 9 | 38.1 (29.37) | 35.8 (24.48)
  Hour 12 | 43.6 (33.33) | 38.9 (25.87)
  Hour 18 | 44.5 (29.46) | 50.7 (30.59)
  Hour 24 | 49.3 (32.63) | 40.3 (26.04)
  Hour 36 | 47.0 (32.11) | 27.8 (20.27)
  Hour 48 | 34.2 (27.31) | 27.9 (19.67)
  Hour 72 | 27.4 (24.79) | 34.6 (30.00)
  Hour 96 | 27.1 (23.70) | 19.1 (28.24)

7. Secondary Outcome: VAS (mm) Pain Intensity Scores Over Time (After Cough)
Description: For the VAS assessment, patients measured their pain intensity after aggravated movement (cough) using a horizontal 100-mm VAS scale labeled as follows: No Pain (0 mm) as the left anchor and Worst Pain Imaginable (100 mm) as the right anchor.
Time Frame: Hour 1, 1.5, 2,3,6,9,12,18,24,36,48,72,96
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System
Number analyzed (Participants) | 14 | 13
units on a scale
  Hour 1 | 84.4 (21.41) | 86.1 (21.72)
  Hour 1.5 | 76.5 (24.54) | 79.8 (25.33)
  Hour 2.0 | 73.8 (26.25) | 84.6 (24.19)
  Hour 3.0 | 62.1 (26.52) | 77.1 (31.40)
  hour 6.0 | 61.9 (33.51) | 65.8 (28.50)
  Hour 9.0 | 51.5 (33.07) | 52.5 (28.08)
  Hour 12 | 43.6 (33.33) | 38.9 (25.87)
  Hour 18 | 44.5 (29.46) | 50.7 (30.59)
  Hour 24 | 49.3 (32.63) | 40.3 (26.04)
  Hour 36 | 47.0 (32.11) | 27.8 (20.27)
  Hour 48 | 34.2 (27.31) | 27.9 (19.67)
  Hour 72 | 27.4 (24.79) | 34.6 (30.00)
  Hour 96 | 27.1 (23.70) | 19.1 (28.24)

ADVERSE EVENTS:
Time Frame: Information regarding AEs was collected from the time of hospital admission through Day 30. Normal postoperative sequelae were not considered to be AEs unless they occurred in a more severe form, as judged by the Investigator. Information on AEs was also collected during the Day 8 and Day 30 follow-up calls.
Arm/Group | Bupivacaine Collagen Sponge | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 7/14 | 9/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine Collagen Sponge (N=14) | ON-ON-Q PainBuster Post-op Pain Relief SystemQ System (N=13)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No